CLINICAL TRIAL: NCT07326046
Title: Adolescent Elite Athletes: A Comparative Biomechanical Study of Trunk Mobility, Lower Extremity Flexibility, and Functional Balance Across Sports Branches
Brief Title: Elite Athletes: Trunk Mobility, Lower Extremity Flexibility, and Functional Balance Across Sports
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Other Study IDs: TEF-BALANCE
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain
Keywords: Dynamic Q Angle; ore Endurance; Lower Extremity Function; Adolescent Athletes
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PFPS Group/ Cohort: Adolescent elite athletes diagnosed with patellofemoral pain syndrome.
- Control Group: Healthy adolescent elite athletes without anterior knee pain or lower extremity complaints.

SUMMARY:
This cross-sectional observational study investigated the relationships among dynamic Q angle, core muscle endurance, hip flexibility, and lower extremity functional status in elite adolescent athletes with and without patellofemoral pain syndrome (PFPS). A total of 75 track-and-field athletes aged 15-18 years were included, 42 with PFPS and 33 healthy controls. Dynamic Q angle was assessed using a digital goniometric analysis of the step-down test, core endurance was measured with the McGill endurance tests, flexibility was evaluated using the Straight Leg Raise, Modified Thomas, and Ober tests, and functional status was assessed with the Lower Extremity Functional Scale (LEFS).

The study found that athletes with PFPS demonstrated a higher dynamic Q angle, lower core extension and lateral endurance, reduced hip flexor and iliotibial band flexibility, and lower functional scores compared with controls. Regression analyses indicated that hip flexor tightness and functional capacity were significant predictors of the dynamic Q angle in the PFPS group. These findings suggest that PFPS in adolescent athletes is a multidimensional condition influenced by proximal endurance, flexibility, and dynamic alignment rather than isolated knee-level factors.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is a common overuse condition in adolescent athletes and is associated with pain, performance limitations, and reduced participation in sports activities. Increasing evidence suggests that PFPS is not limited to local knee pathology, but is influenced by proximal neuromuscular control, dynamic alignment, and soft-tissue flexibility. The dynamic Q angle, which reflects frontal-plane knee alignment during functional tasks, has been proposed as a clinically meaningful indicator of patellofemoral loading; however, the interaction between dynamic alignment, core endurance, and flexibility parameters in adolescent elite athletes remains insufficiently explored.

This cross-sectional observational study was conducted to examine the relationships among dynamic Q angle, core muscle endurance, hip and lower extremity flexibility, and functional status in elite adolescent athletes with and without PFPS. A total of 75 track-and-field athletes aged 15-18 years were included. Participants were allocated into two groups: athletes diagnosed with PFPS and healthy controls. Dynamic Q angle was assessed using digital two-dimensional video analysis of the step-down test. Core endurance was evaluated using the McGill endurance test battery (flexor, extensor, and lateral plank tests). Flexibility was assessed using the Straight Leg Raise, Modified Thomas, and Ober tests. Functional status was measured with the Lower Extremity Functional Scale (LEFS). All side-dependent measurements were analyzed on the index limb (symptomatic side in the PFPS group and matched limb in controls).

Group differences and correlations among variables were examined, and multiple regression analyses were performed to identify predictors of the dynamic Q angle. The results demonstrated that athletes with PFPS exhibited a significantly higher dynamic Q angle, reduced core extension and lateral endurance, decreased hip flexor and iliotibial band flexibility, and lower functional scores compared with controls. In the PFPS group, hip flexor tightness and functional capacity were significant predictors of the dynamic Q angle, explaining a substantial proportion of its variance.

These findings indicate that PFPS in adolescent athletes represents a multidimensional biomechanical syndrome characterized by the interaction of proximal stability, flexibility restrictions, and dynamic alignment alterations. The study highlights the clinical importance of comprehensive assessment strategies that incorporate core endurance, hip flexibility, and functional performance measures, rather than focusing solely on isolated knee-level factors. The results may contribute to the development of targeted prevention and rehabilitation strategies for adolescent athletes at risk of PFPS.

ELIGIBILITY:
Inclusion Criteria:

* Elite adolescent track-and-field athletes aged 15-18 years
* Minimum 2 years of regular training participation
* Training at least 5 days per week
* Ability to complete all assessment procedures
* PFPS group: history of anterior knee pain associated with activity, positive clinical provocation tests, and AKPS score < 80
* Control group: no history of lower extremity pain or functional limitation

Exclusion Criteria:

* History of lower extremity surgery or acute injury within the past 6 months
* Neurological, rheumatological, or systemic disease
* Structural deformity of the hip, knee, or ankle
* Ongoing orthopedic rehabilitation or regular analgesic / anti-inflammatory medication use
* Any condition preventing participation in the tests or introducing measurement bias

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Elite adolescent track-and-field athletes training within national athletic development programs.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Dynamic Q Angle | Single assessment at baseline (cross-sectional).
  Dynamic Q angle measured on the index limb during the step-down test using 2-dimensional digital goniometric video analysis. Higher values indicate greater frontal-plane malalignment.
Core Muscle Endurance - Extension Test | Single assessment at baseline.
  Duration (seconds) of trunk extensor endurance test from the McGill protocol. Longer duration reflects better endurance capacity.
Hip Flexor Flexibility - Modified Thomas Test | Baseline, single assessment.
  Hip flexion angle obtained during the Modified Thomas test on the index limb. Greater angles indicate muscle tightness.
Core Muscle Endurance - Lateral Plank Test | Single assessment at baseline.
  Duration (seconds) of lateral plank endurance on the index limb according to the McGill protocol.
Iliotibial Band / TFL Flexibility - Ober Test | Baseline, single assessment.
  Adduction angle recorded during the Ober test on the index limb. Lower adduction indicates greater tightness.
Hamstring Flexibility - Straight Leg Raise Test | Single assessment at baseline.
  Hip flexion angle at the onset of pelvic compensation during passive straight leg raise. Higher angles reflect better flexibility.
Functional Status - Lower Extremity Functional Scale (LEFS) | Baseline, single assessment.
  Self-reported lower-limb functional capacity scored from 0-80, with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Locations (1):
- Burcin Ugur Tosun, Famagusta, Cyprus